CLINICAL TRIAL: NCT00312195
Title: An Open-label Run-in, Followed by a Randomized, Double-blind, Placebo Controlled, Parallel Group Study to Show the Effectiveness of Buprenorphine Transdermal System in Management of Patients With Chronic Nonmalignant Pain Syndromes
Brief Title: Safety and Efficacy of Buprenorphine Transdermal System (BTDS) in Subjects With Chronic Nonmalignant Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Collaborators: Napp Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BUP3201
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Results first posted 2010-10-15 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Non-malignant Pain
Keywords: Chronic pain; opioid; transdermal; Butrans™ [BTDS]
MeSH Terms: conditions — Chronic Pain | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- BTDS (5, 10 or 20) (Experimental): Buprenorphine transdermal patch
  Interventions: Drug: Buprenorphine transdermal patch
- Placebo to match BTDS (Placebo Comparator): Placebo to match buprenorphine transdermal patch
  Interventions: Drug: Placebo to match BTDS

INTERVENTIONS:
Drug: Buprenorphine transdermal patch — Buprenorphine transdermal patch 5, 10 or 20 mcg/h applied for 7-day wear.
  Other Names: Butrans™
  Arms: BTDS (5, 10 or 20)
Drug: Placebo to match BTDS — Placebo to match buprenorphine transdermal patch applied for 7-day wear.
  Arms: Placebo to match BTDS

SUMMARY:
The objective of this study is to demonstrate the effectiveness and tolerability of the buprenorphine transdermal system (5, 10 and 20) in comparison to matching placebo transdermal system in subjects with chronic nonmalignant pain syndromes currently controlled by oral opioids. The double-blind treatment intervention duration is 2 weeks during which time supplemental analgesic medication (acetaminophen) will be provided to all subjects in addition to study drug.

DETAILED DESCRIPTION:
Buprenorphine is a synthetic opioid analgesic with over 25 years of international clinical experience indicating it to be safe and effective in a variety of therapeutic situations for the relief of moderate to severe pain.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 month's history of nonmalignant pain, currently in stable pain control on opioid therapy.
* Good, very good or excellent pain control on current opioid therapy.
* Willing and able to use a telephone interactive voice response service.

Exclusion Criteria:

* Currently receiving daily morphine or oxycodone monotherapy.
* Scheduled for surgery of the disease site (eg, major joint replacement surgery), or any other major surgery, which would fall within the study period.

Other protocol-specific exclusion/inclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2001-03; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (42):
- United States (21):
  - Hawthorne and York, Phoenix, Arizona
  - Arizona Research Center Inc, Phoenix, Arizona
  - Clinical Research Consultants Inc, Trumbull, Connecticut
  - Tampa Bay Medical Research Inc, Clearwater, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - University Clinical Research Deland, DeLand, Florida
  - University Clinical Research Inc,, Pembroke Pines, Florida
  - Gold Coast Research LLC, Plantation, Florida
  - Gold Coast Research LLC, Tamarac, Florida
  - Family Medicine Associates, Evansville, Indiana
  - Pain Management and Rehabilitation, Terre Haute, Indiana
  - Southeastern Center for Headache and Pain, Crestview Heights, Kentucky
  - Westside Family Medical Center PC, Kalamazoo, Michigan
  - The Arthritis Clinic, Charlotte, North Carolina
  - Cornerstone Research Care, High Point, North Carolina
  - ALL-TRIALS Clinical Research LLC, Winston-Salem, North Carolina
  - Private Practice, Chardon, Ohio
  - Summit Research Solutions, Memphis, Tennessee
  - Radiant Research, Austin, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Clinical Research Management, New Berlin, Wisconsin
- United Kingdom (21):
  - Whiteabbey Health Centre, Newtownabbey, Belfast
  - Antrim Coast Fundholding Group, Lame, Co Antrim
  - Portglenone Health Centre, Portglenone, CO Antrim
  - Garden Street Surgery, Magherafelt, Co Derry
  - Springhill Surgery, Bangor, Co Down
  - Bennett Road Surgery, Keresley End, Coventry
  - Little Common Surgery, Bexhill-on-Sea, E Sussex
  - Old Town Surgery, Bexhill-on-Sea, E Sussex
  - Roebuck House Surgery, Hastings, E Sussex
  - Leslie Surgery, Glenrothes, Fife
  - Valleyfield Health Centre, High Valleyfield, Fife
  - Townhead Health Centre, Glasgow, Glasgow
  - Castlemilk Health Centre, Glasgow, Glasgow
  - Ashvale Health Centre, Aldershot, Hants
  - The Academy Medical Practice, Coatbridge, Lanarkshire
  - Sanbury Health Centre Group Practice, Sunbury-on-Thames, Middx
  - Houston Surgery, Houston, Renfrewshire
  - The Burns Practice, Doncaster, S Yorkshire
  - Grosvenor Medical Centre, Royal Tunbridge Wells, W Sussex
  - Gables Medical Section, Coventry, Warwickshire
  - The Ridge Medical Practice, Great Horton, Bradford, West Yorkshire

RESULTS

PARTICIPANT FLOW:
Recruitment Details: (First patient first visit) 19-Mar-2001 to (last patient last visit) 22-Jul-2001 at 42 centers: 21 in the UK and 21 in the US.
Pre-assignment Details: The Run-in period (N = 588 subjects started) consisted of titration from buprenorphine transdermal patch (BTDS) 5 to BTDS 10, or 20 mcg/h for tolerability. If BTDS was not tolerated or pain increased, the subject was discontinued. N = 267 subjects were randomized.
Groups:
- Double-blind Placebo Patch: Reference drug - Placebo transdermal patch to match BTDS 5, 10, or 20 mcg/h applied for 7-day wear.
- Double-blind BTDS: Test drug - buprenorphine transdermal patch (BTDS) 5, 10, or 20 mcg/h applied for 7-day wear.
Period: Overall Study
Arm/Group | Double-blind Placebo Patch | Double-blind BTDS
Started | 138 | 129
Completed | 132 | 123
Not Completed | 6 | 6
Not completed — Adverse Event | 4 | 6
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind Placebo Patch | Double-blind BTDS | Total
Number analyzed (Participants) | 138 | 129 | 267
Age Continuous [Mean (Standard Deviation); unit: years] | 59.2 (11.48) | 56.2 (13.34) | 57.7 (12.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 79 | 167
  Male | 50 | 50 | 100
Region of Enrollment [Number; unit: participants]
  United States | 46 | 42 | 88
  United Kingdom | 92 | 87 | 179

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects With Ineffective Treatment During the Double-blind Evaluation Phase.
Description: Ineffective treatment was defined as:
  * Subject took >1 gram of acetaminophen in a 24-hour period, or
  * Subject required a change in transdermal patch (TDS) dose, or
  * Subject had difficulty in keeping the TDS on, or
  * Subject discontinued due to ineffective treatment (but did not meet any of the above criteria).
  Note: some subjects may have had multiple reasons for ineffective treatment and are counted under each category. Therefore the sum of subjects across all criteria for ineffective treatment is greater than the total number of subjects with ineffective treatment.
Time Frame: Double-blind phase (14 days)
Population: The Full Analysis Population (N = 266) for efficacy analyses included all subjects who were randomized and provided at least 1 efficacy assessment in the double-blind phase.
Measure: Number; unit: participants
Groups:
- Double-blind BTDS: Test drug - buprenorphine transdermal patch 5, 10 or 20 mcg/h applied for 7-day wear.
- Total: Placebo and BTDS combined.
Arm/Group | Double-blind Placebo Patch | Double-blind BTDS | Total
Number analyzed (Participants) | 137 | 129 | 266
participants
  Subjects With Ineffective Treatment | 89 | 66 | 155
  Reason: took more than 1 gram of acetaminophen/day | 81 | 59 | 140
  Reason: required a change in TDS dose | 34 | 25 | 59
  Reason: difficulty keeping patch on | 6 | 1 | 7
  Reason: discontinued due to ineffective treatment | 2 | 3 | 5
Statistical Analysis 1: Comparison: Double-blind Placebo Patch vs Double-blind BTDS; H0: the odds of ineffective treatment is the same for subjects receiving placebo as for those receiving BTDS versus the alternative H1: the odds of ineffective treatment is different for subjects receiving placebo from those receiving BTDS; Test type: Superiority or Other; p = .0217, Regression, Logistic — P value is from a logistic regression analysis with terms for treatment effect, country and pain site (hip, knee, back and other); Odds Ratio (OR) = 1.79, 95% CI 2-sided [1.09 to 2.95], Standard Error of Mean .2544 — Primary variable was defined as: ratio of the probability of having ineffective treatment divided by the probability of having effective treatment

2. Secondary Outcome: Time (Days) From the Initial Dose of Study Drug in the Double-blind Evaluation Phase to Ineffective Treatment
Description: The time of ineffective treatment was calculated as the earliest of the following:
  * The date the subject first took >1 gram of acetaminophen,
  * The visit date when ineffective treatment was first determined, or
  * The date the last patch was removed.
Time Frame: 14 days
Population: Full Analysis (N = 266) consisted of subjects who were randomized into the double-blind evaluation phase, were exposed to study drug, and provided at least 1 efficacy assessment during the double-blind evaluation phase.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Double-blind Placebo Patch | Double-blind BTDS
Number analyzed (Participants) | 137 | 129
Days | 5.6 (0.44) | 7.4 (0.45)

3. Secondary Outcome: The Number of Subjects Who Had Ineffective Treatment or Who Discontinued Due to Reasons Other Than Ineffective Treatment in the Double-blind Phase
Description: Note: The total numbers of "Subjects w/ineffective treatment or who discont'd" for placebo and BTDS are 1 less because there were reasons other than lack of efficacy that made up this total: adverse event, death, lost to follow- up, protocol violation, and other. Example for placebo 89+5=94; however, 93 is indicated for the total because there is 1 subject in the placebo group who was counted under ineffective treatment and discontinued due to reasons other than lack of efficacy. The same is true for 1 subject in BTDS.
Time Frame: 14 days
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Double-blind Placebo Patch | Double-blind BTDS
Number analyzed (Participants) | 137 | 129
participants
  Subjects w/ineffective treatment or who discont'd | 93 | 71
  Ineffective Treatment | 89 | 66
  Discontinued due to other reasons | 5 | 6

4. Secondary Outcome: The Amount of Rescue Medication Used for Pain (Average Daily Number of Acetaminophen Tablets).
Description: The average daily acetaminophen (Panadol) use (1 tablet = 500 mg) during the double-blind phase was compared between the treatment groups using ANCOVA methodology with terms for country and treatment. The average escape medication used in the last 4 days prior to randomization was included as a covariate.
Time Frame: 14 days
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Tablets
Arm/Group | Double-blind Placebo Patch | Double-blind BTDS
Number analyzed (Participants) | 137 | 129
Tablets | 2.2 (0.15) | 1.8 (0.14)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs)that occurred after the signing of the informed consent up to end of study, discontinuation, or Serious AE occurring up to 30 days following the last study visit were followed until the AE resolved.
Description: Adverse Events were learned of through spontaneous reports and subject interview.
Groups:
- Open-label Run-in Period BTDS 5, 10 or 20: Buprenorphine transdermal patch (BTDS) 5, 10, or 20 mcg/h applied for 7-day wear.
Arm/Group | Double-blind Placebo Patch | Double-blind BTDS | Open-label Run-in Period BTDS 5, 10 or 20
Serious Adverse Events (participants affected / at risk) | 0/138 | 0/129 | 7/588
Other Adverse Events (participants affected / at risk) | 21/138 | 25/129 | 245/588
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Placebo Patch (N=138) | Double-blind BTDS (N=129) | Open-label Run-in Period BTDS 5, 10 or 20 (N=588)
Pain abdominal (General disorders) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Abscess (General disorders) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Injury accidental (General disorders) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Cellulitis (General disorders) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Pain, chest (General disorders) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Fibrillation, atrial (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Gastroenteritis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) — Systematic and nonsystematic assessments
Depression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
OTHER ADVERSE EVENTS (reported when occurring in more than 4.50% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo Patch (N=138) | Double-blind BTDS (N=129) | Open-label Run-in Period BTDS 5, 10 or 20 (N=588)
Headache (General disorders) | 3 | 5 | 44 — Systematic and nonsystematic assessments
Asthenia (General disorders) | 3 | 2 | 36 — Systematic and nonsystematic assessments
Nausea (Gastrointestinal disorders) | 5 | 4 | 112 — Systematic and nonsystematic assessments
Vomit (Gastrointestinal disorders) | 0 | 1 | 36 — Systematic and nonsystematic assessments
Dizziness (Nervous system disorders) | 0 | 0 | 73 — Systematic and nonsystematic assessments
Somnolence (Nervous system disorders) | 1 | 3 | 41 — Systematic and nonsystematic assessments
Erythema at site (Skin and subcutaneous tissue disorders) | 18 | 17 | 43 — Systematic and nonsystematic assessments
Pruritus at site (Skin and subcutaneous tissue disorders) | 7 | 12 | 58 — Systematic and nonsystematic assessments

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days